CLINICAL TRIAL: NCT04656262
Title: The METROPHOLYS Study Metronomic Cyclophosphamide vs Doxorubicin in Elderly Patients With Advanced Soft Tissue Sarcomas Randomized, Controlled Open Label Clinical Trial
Brief Title: Low Dose Continuous Cyclophosphamide vs Standard Doxorubicin in Advanced Sarcoma Elderly Patients
Acronym: METROPHOLYS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: enrollment too slow to reach the target in a reasonable time frame
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-2018-STS-METROPHOLYS
Record Dates: First submitted 2020-11-25; First posted 2020-12-07 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Soft Tissue Sarcoma Adult
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronomic cyclophosphamide (Experimental): Cyclophosphamide 50 mg daily per os continuously; Patients will be visited for re-cycling every three weeks. Metronomic cyclophosphamide will be taken in the morning along with a full glass of water.
  Interventions: Drug: Cyclophosphamide
- Doxorubicin (Active Comparator): Doxorubicin 60 mg/mq i.v. in 10 minutes, day 1; to be repeated every three weeks up to a maximum of 6 cycles.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide is formulated as coated tablets of 50mg for oral administration
  Other Names: Endoxan
  Arms: Metronomic cyclophosphamide
Drug: Doxorubicin — Doxorubicin is formulated as 60 mg/mq for infusional use (i.v use)
  Arms: Doxorubicin

SUMMARY:
To compare the efficacy, as measured by time to treatment failure, of metronomic cyclophosphamide with respect to doxorubicin in elderly patients affected by mSTS.

DETAILED DESCRIPTION:
This phase III randomized clinical trial was designed to compare metronomic Cyclophosphamide with standard Doxorubicin for the first-line treatment of elderly cancer patients with advanced inoperable or metastatic STS:

i) ARM A (experimental): Metronomic Cyclophosphamide ii) ARM B (control): Doxorubicin up to six cycles

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all the following criteria:

1. Histologically proven diagnosis of soft tissue sarcoma.
2. Advanced unresectable or metastatic soft tissue sarcoma not previously treated with chemotherapy for metastatic disease.
3. At least one measurable lesion according to RECIST1.1 criteria.
4. Availability of a tumor sample (primary and/or metastatic sites).
5. Age ≥ 70 years (70-75 years if UNFIT at G8; >75 independent of G8 score)
6. ECOG PS 0-2.
7. Life expectancy of at least 12 weeks.
8. Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hgb ≥ 9 g/dl.
9. Adequate hepatic function, defined as: Total bilirubin ≤ 1.5 time the upper-normal limits (ULN) of the normal values, ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 x ULN (or <5 x ULN in case of liver metastases)
10. Alkaline phosphatase ≤ 2.5 x ULN (or <5 x ULN in case of liver metastases).
11. Creatinine clearance ≥ 30 mL/min.
12. Normal cardiac function, with left ventricular ejection fraction (LVEF) ≥50%.
13. Male subjects with female partners of childbearing potential must be willing to use adequate contraception as approved by the investigator
14. Geriatric assessment by means of G8 screening tool and CRASH score.
15. Will and ability to comply with the protocol.
16. Written informed consent to study participation.

Exclusion Criteria:

* Patients will be excluded from the study for any of the following reasons:

  1. Previous treatment for metastatic disease.
  2. Previous (neo) adjuvant chemotherapy with anthracyclines.
  3. Radiotherapy to any site within 4 weeks before the study.
  4. Untreated brain metastases or spinal cord compression or primary brain tumors.
  5. Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration.
  6. Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), serious cardiac arrhythmia requiring medication.
  7. Treatment with any investigational drug within 30 days prior to enrollment or 2 investigational agent half-lives (whichever is longer)
  8. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ.
  9. Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
  10. Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.
  11. Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.
  12. Sexually active males unwilling to practice contraception during the study and until 6 months after the last trial treatment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | From date of randomization until the date of treatment discontinuation due to disease progression, toxicity leading to treatment discontinuation, or death, whichever occurs first, assessed up to 12 months
  Progressive disease is defined as per RECIST 1.1 criteria based on investigator assessment.
  Toxicity is assessed according to NCI-CTCAE criteria v. 4.03

SECONDARY OUTCOMES:
Progression free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progressive disease is defined as per RECIST 1.1 criteria based on investigator assessment.
Overall survival | Time from randomization to the date of death due to any cause or last follow up assessed up to 12 months
  Overall Survival is defined as the time from date of randomization to the date of death due to any cause
Overall Toxicity Rate | From signing IC until 30 days after last study treatment
  Toxicities will be recorded, classified, graded and managed according to NCI CTCAE v. 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Brunello, Principal Investigator — Istituto Oncologico Veneto
Locations (13):
- Italy (13):
  - Policlinico Sant'Orsola Malpighi, Bologna, BO
  - Istituto Clinico Humanitas, Rozzano, MI
  - Istituto Ortopedico Rizzoli IRCCS, Bologna
  - Fondazione del Piemonte per l'Oncologia IRCCS, Candiolo
  - IRST Romagnolo IRCCS, Meldola
  - Istituto Nazionale Tumori IRCCS, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
  - AOU Policlinico Giaccone Palermo, Palermo
  - Ospedale Misericordia e Dolce, Prato
  - Policlinico Universitario Campus Biomedico, Roma
  - IFO - Istituto Regina Elena, Roma
  - Presidio Sanitario Humanitas - Gradenico, Torino
  - AOUI Policlinico Borgo Roma, Verona